CLINICAL TRIAL: NCT00751569
Title: microRNA Profile in Umbilical Cord Blood NK Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-Wu Lin, national Taiwan University Hospital
Other Study IDs: 200808006R
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Pregnant Women
Keywords: umbilical cord blood
MeSH Terms: interventions — Blood Donation

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Umbilical cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A1: A group of 3 to 5 pregnant women as donors for umbilical cord blood
  Interventions: Other: blood donation

INTERVENTIONS:
Other: blood donation — obtaining cord blood
  Other Names: cord blood donation

SUMMARY:
Umbilical cords contain immature blood cells, including a group of lymphocytes, that are important in the so-called natural immunity. We want to study the cytokine levels in umbilical cord NK cells and its regulation a family of newly identified small RNAs (microRNAs).

DETAILED DESCRIPTION:
Our preliminary data pointed to the possibility of cytokine regulation by microRNAs in NK lymphoma and NK lymphoma cell lines. We want to use umbilical cord blood as controls for the biological significance in normal NK cell development.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnant women

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: normal pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2008-09; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Wu Lin, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan